CLINICAL TRIAL: NCT01400568
Title: A Methodological Pilot Study to Assess the Suitability of a Low Dose LPS Inhalation as a Challenge Model in Early Translational Drug Development
Brief Title: Suitability of a Low Dose Lipopolysaccharide (LPS) Inhalation as a Challenge Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Prof. Dr. Jens Hohlfeld, Fraunhofer ITEM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-06 LOPS
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LPS challenge and fluticasone propionate (Experimental): In case LPS induced airway inflammation is reproducible, the effect of a single high dose of inhaled fluticasone propionate will be assessed after a 4-week wash-out period.
  Interventions: Drug: LPS challenge with nebulized LPS; Drug: fluticasone propionate (FP)

INTERVENTIONS:
Drug: LPS challenge with nebulized LPS — 20,000 EU of Clinical Center Reference Endotoxine (CCRE) will be applied by an AKITA® Jet Nebulizer under the constant supervision of the site staff.
Drug: fluticasone propionate (FP) — The dosage of FP will be 2 mg. This dosage will be inhaled by 4 puffs of Flutide® forte 500 Diskus® 500 µg / dose according to the package insert.

SUMMARY:
This pilot study is planned to assess the suitability of a low dose Lipopolysaccharide (LPS) inhalation as a challenge model. As LPS effects are based on a different mode of action, this challenge model will provide the possibility to test a wider spectrum of potential drugs in the future. Provided that the LPS response is reproducible, it is planned to test whether a single high dose of inhaled steroid can serve as a positive control in the LPS model. Another major aim of the study is to test a variety of novel tools for the non-invasive assessment of airway inflammation induced by LPS challenge.

DETAILED DESCRIPTION:
In this study, airway inflammation will be induced by LPS inhalation. In case a neutrophilic airway inflammation can be safely induced by inhaled LPS, the LPS challenge will be repeated. If neutrophil airway inflammation after LPS challenge is reproducible LPS challenge will be repeated after pre-treatment with a single high dose of inhaled fluticasone propionate.

To determine airway inflammation, the subjects' exhaled breath will be analyzed by different techniques, and blood samples as well as induced sputum will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Healthy male and female nonsmokers, aged 18 to 55 years, with a history of less than 1 pack year having been nonsmokers for at least the last five years
* FEV1 ≥ 80 % of predicted, FEV1/FVC ≥ 70 %.
* Available to complete all study measurements
* Subjects must be able to produce adequate sputum (≥ 1× 106 total cells, ≥ 50 % cell viability, ≤ 20 % squamous epithelial cells)
* Negative methacholine challenge (> 8 mg/mL)
* Women will be considered for inclusion if they are:

Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).

Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

Exclusion Criteria:

* Upper or lower respiratory tract infection in the last four weeks prior to screening
* Past or present disease, which as judged by the investigator, may affect the outcome of the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
* Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
* Administration of corticosteroids within the last 2 weeks prior to screening. Administration of topical corticosteroids within the last 2 weeks prior to screening is permitted at the discretion of the investigator.
* History of drug or alcohol abuse
* Risk of non-compliance with study procedures
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Induced sputum | 6 h after the start of LPS challenge
  • neutrophil cell count

SECONDARY OUTCOMES:
lung function | at the end of each LPS challenge and up to 24 hours
  Change of lung function directly at the end of each challenge as well as up to 24 h after the end of exposure compared with baseline
Blood samples | before and 6 h after the start of LPS challenge
  Differential cell count
Exhaled breath | 3 hours after the start of LPS challenge
  Pre-concentrated samples (30 L, 10-15 exhalations) on a specific substrate for later analysis by Gas Chromatorgraphy - Mass Spectrometry (GC-MS) or Smart-Nose and exhaled breath temperature
Induced sputum | 6 h after the start of LPS challenge
  soluble biomarkers such as but not limited to Myeloperioxidase (MPO), Surfactant Protein D (SP-D), Interleukin (IL-8)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Professor, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Janssen O, Schaumann F, Holz O, Lavae-Mokhtari B, Welker L, Winkler C, Biller H, Krug N, Hohlfeld JM. Low-dose endotoxin inhalation in healthy volunteers--a challenge model for early clinical drug development. BMC Pulm Med. 2013 Mar 28;13:19. doi: 10.1186/1471-2466-13-19. PMID 23537365